CLINICAL TRIAL: NCT04318678
Title: CD123-Directed T-Cell Therapy for Acute Myelogenous Leukemia (CATCHAML)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CATCHAML
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: AML/MDS; B-ALL; T-ALL; BPDCN
Keywords: CD123+
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Blastic Plasmacytoid Dendritic Cell Neoplasm | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Mesna; Rituximab

STUDY DESIGN:
Intervention Model Description: Due to review of dose limiting toxicity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARM A CD123-CAR T cell therapy (Other): For patients who have not received an allogeneic transplant or for patients who have received allogeneic transplant and do not have a transplant donor available
  CD123-CAR T-cell dose and infusion Up to 4 Dose levels will be evaluated with a maximum dose of 2.5 x 10^8 CAR+ T cells. If dose limiting toxicities (DLTs) are observed on Dose level 1 then the cell dose is de- escalated.
  Interventions: Drug: CD123-CAR T; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna; Drug: Rituximab
- ARM B CD123-CAR T cell therapy (Experimental): For patients who relapsed following allogeneic transplant and whose CAR T-cells will be manufactured from the previous transplant donor, when available.
  CD123-CAR T-cell dose and infusion Up to 4 Dose levels will be evaluated with a maximum dose of 2.5 x 10^8 CAR+ T cells. If dose limiting toxicities (DLTs) are observed on Dose level 1 then the cell dose is de- escalated.
  Interventions: Drug: CD123-CAR T; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna; Drug: Rituximab

INTERVENTIONS:
Drug: CD123-CAR T — To treat relapsed/refractory CD123+ AML/MDS, B-ALL, T-ALL or BPDCN patient population that needs new cancer-directed therapies.
  Other Names: CD123-CAR T cells
Drug: Cyclophosphamide — Cyclophosphamide is a nitrogen mustard derivative. It acts as an alkylating agent that causes cross-linking of DNA strands by binding with nucleic acids and other intracellular structures, thus interfering with the normal function of DNA.
  Other Names: Cytoxan
Drug: Fludarabine — Fludarabine phosphate is a synthetic purine nucleoside analog. It acts by inhibiting DNA polymerase, ribonucleotide reductase and DNA primase by competing with the physiologic substrate, deoxyadenosine triphosphate, resulting in inhibition of DNA synthesis
  Other Names: Fludara
Drug: Mesna — Mesna is a synthetic sulfhydryl (thiol) compound. Mesna contains free sulfhydryl groups that interact chemically with urotoxic metabolites of oxaza-phosphorine derivatives such as cyclophosphamide and ifosfamide
Drug: Rituximab — Rituximab is a monoclonal antibody directed against the CD20 antigen on the surface of B-lymphocytes
  Other Names: Rituxan

SUMMARY:
The CD123-CAR T-cell therapy is a new treatment that is being investigated for treatment of AML/myelodysplastic syndrome (MDS), T- or B- acute lymphoblastic leukemia (ALL) or blastic plasmacytoid dendritic cell neoplasia (BPDCN). The purpose of this study is to find the maximum (highest) dose of CD123-CAR T cells that is safe to give to these patients. This would include studying the side effects of the chemotherapy, as well as the CD123-CAR T-cell product on the recipient's body, disease and overall survival.

Primary Objective:

* To determine the safety of one intravenous infusion of escalating doses of autologous, CD123-CAR T cells in patients (≤21 years) with recurrent/refractory CD123+ disease (AML/MDS, B-ALL, T-ALL or BPDCN) after lymphodepleting chemotherapy.
* To determine the safety of an intravenous infusion of escalating doses of donor derived, CD123-CAR T cells in patients (≤21 years) with recurrent/refractory CD123+ disease (AML/MDS, B-ALL, T-ALL, BPDCN or MPAL) after lymphodepleting chemotherapy.

Secondary Objectives

- To evaluate the antileukemia activity of CD123-CAR T cells.

Exploratory Objectives

* To assess the immunophenotype, clonal structure and endogenous repertoire of CD123-CAR T cells and unmodified T cells
* To characterize the cytokine profile in the peripheral blood and CSF after treatment with CD123-CAR T cells
* To characterize tumor cells post CD123-CAR T-cell therapy
* To compare in vivo properties of donor-derived versus autologous CD123- CAR T cells

DETAILED DESCRIPTION:
This study will evaluate the safety and maximum tolerated dose of CD123-CAR T cells.

This study contains 2 phases. The first part is the called the "Collection and Manufacturing Phase" and the second is the "Treatment Phase".

The Collection and Manufacturing Phase refers to your blood cells being collected and possibly frozen, via a process called apheresis. These cells will then be changed to improve their ability to recognize and kill cancer cells.

The Treatment Phase refers to the portion of the study in which you receive an infusion of the CD123-CAR T cells that were made in the Collection and Manufacturing Phase; chemotherapy is given for several days prior to the cellular infusion. You are then monitored for any possible side effects.

.

Chemotherapy is given to get your body ready to accept the CATCHAML treatment.

Treatment Schedule:

Patients will receive lymphodepleting chemotherapy followed by infusion of CD123-CAR T cells

Fludarabine on day -4, -3 and -2

Cyclophosphamide on day -3 and -2

REST DAY on day -1

CD123-CAR T cell infusion on day 0 or +1

ELIGIBILITY:
Inclusion Criteria for Procurement and T-cell Production:

* Age ≤21 years old
* Relapsed/refractory CD123+ disease defined as follows:

AML/MDS

* Relapsed disease: Patients developing recurrent disease after a first complete remission (CR)
* Refractory disease: Patients not achieving a CR after 2 cycles of induction chemotherapy

B-cell ALL

* Relapsed disease that is CD123 positive and CD19 negative/dim or patients otherwise ineligible for CD19 directed therapies including

  * Patients in 2nd or greater relapse
  * Patients with relapse after allogeneic HSCT
* Refractory disease that is CD123 positive and CD19 negative/dim or patients otherwise ineligible for CD19 directed therapies

T-cell All • Relapsed refractory disease that is CD123 positive

BPDCN

• Relapsed/refractory disease that has failed front-line therapy

* Estimated life expectancy of >12 weeks
* Karnofsky or Lansky (age-dependent) performance score ≥50
* Patients with a history of prior allogeneic HCT must be clinically recovered from prior HCT therapy, have no evidence of active GVHD and have not received a donor lymphocyte infusion (DLI) within the 28 days prior to apheresis
* Patient must have an identified, suitable HCT donor
* For females of child-bearing age:
* Not lactating with intent to breastfeed
* Not pregnant with negative serum pregnancy test within 7 days prior to enrollment
* Meets eligibility criteria to undergo autologous apheresis, or have previously undergone autologous apheresis

Exclusion Criteria:

* Known primary immunodeficiency
* History of HIV infection
* Severe intercurrent uncontrolled bacterial, viral or fungal infection (e.g. active hepatitis B or C infection or adenovirus infection)
* History of hypersensitivity reactions to murine protein-containing products
* Patients with acute promyelocytic leukemia (APL, t (15;17))
* Known contraindication to the protocol defined lymphodepleting chemotherapy regimen of fludarabine/cyclophosphamide.

Inclusion Criteria for Treatment:

* Age≤21 years old
* Detectable disease that is CD123+ (at least MRD+ disease)
* Estimated life expectancy of >8 weeks
* Karnofsky or Lansky (age-dependent) performance score≥50
* Patients with a history of prior allogeneic HCT must be clinically recovered from prior HCT therapy, have no evidence of active GVHD and have not received a donor lymphocyte infusion (DLI) within the 28 days prior to planned infusion
* Patient must have an identified, suitable HCT donor
* Adequate cardiac function defined as left ventricular ejection fraction >40%, OR shortening fraction ≥25%
* EKG without evidence of clinically significant arrhythmia
* Adequate renal function defined as creatinine clearance or radioisotope GFR ≥50 ml/min/1.73m2 (GFR ≥40 ml/min/1.73m2 if < 2 years of age)
* Adequate pulmonary function defined as forced vital capacity (FVC)≥50% of predicted value; or pulse oximetry≥92% on room air if patient is unable to perform pulmonary function testing
* Total Bilirubin≤3 times the upper limit of normal for age, except in subjects with Gilbert's syndrome
* Alanine aminotransferase (ALT) OR aspartate aminotransferase (AST) ≤5 times the upper limit of normal for age
* Has recovered from all NCI CTAE grade III-IV, non-hematologic acute toxicities from prior therapy
* For females of child-bearing age

  * Not lactating with intent to breastfeed
  * Not pregnant with negative serum pregnancy test within 7 days prior to enrollment
* If sexually active, agreement to use birth control until 3 months after T- cell infusion. Male partners should use a condom.
* Available autologous transduced T-cell product that has met GMP release criteria

Exclusion Criteria:

* Known primary immunodeficiency
* History of HIV infection
* Severe intercurrent uncontrolled bacterial, viral or fungal infection
* History of hypersensitivity reactions to murine protein-containing products
* History of severe hypersensitivity reactions to cornstarch or hydroxyethyl starch.
* Receiving systemic steroids therapy exceeding the equivalent of 0.5 mg/kg/day of methylprednisolone, in the 7 days prior to CD123-CAR T- cell infusion
* Receiving systemic therapy in the 14 days prior to CD123-CAR T-cell infusion, which will interfere with the activity of the CD123-CAR T cells in vivo (in the opinion of the study PI(s))
* Receiving rituximab therapy in the 30 days prior to CD123-CAR T cell infusion. (This exclusion criterion is intended to prevent premature exposure of CD123-CAR T cells to rituximab, which would activate the safety switch and promote CAR T-cell apoptosis).
* Receiving intrathecal chemotherapy in the 7 days prior to CD123-CAR T cell infusion.
* Known contraindication to the protocol defined lymphodepleting chemotherapy regimen of fludarabine/cyclophosphamide.
* Active CNS disease

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2029-07-29 (Estimated); Study Completion 2030-07-29 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of CD123-CAR T cells (CATCHAML) | 4 weeks after CD123-CAR T-cell infusion
  A phase I design to determine the maximum tolerated dose (MTD) of autologous, CD123- CAR T cells. Four dose levels (3x10^5/kg, 1x10^6/kg, 3x10^6/kg, and 1x10^7/kg) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Swati Naik, MD, Principal Investigator — St. Jude Children's Research Hospital; Paulina Velasquez, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols